CLINICAL TRIAL: NCT02823678
Title: Using Pancreatic Volumetric to Determine the Onset of Diabetes Mellitus and Postoperative Outcomes After Pancreatectomy
Brief Title: Pancreas Volume and Diabetes Status Following Pancreatectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Florida Hospital Tampa Bay Division (Other)
Responsible Party: Principal Investigator, Alexander Rosemurgy, Chief of General Surgery, Florida Hospital Tampa Bay Division
Other Study IDs: 520670
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatectomy: Patients scheduled to undergo a pancreatectomy
  Interventions: Procedure: Pancreatectomy

INTERVENTIONS:
Procedure: Pancreatectomy — Patients will undergo pancreatectomy as part of routine care for their pancreatic neoplasms.

SUMMARY:
This study will enroll 100 patients scheduled to undergo a pancreatectomy.

The primary objective is to develop a scoring system using pancreatic volume measured by CT scan and intraoperative measurements of the pancreas parenchyma to predict the onset of diabetes mellitus after a pancreatectomy. The investigators will also monitor patients with pre-existing diabetes to see if their diabetes worsens or improves.

DETAILED DESCRIPTION:
The primary objective is to develop a scoring system using pancreatic volume measured by CT scan and intraoperative measurements of the pancreas parenchyma to predict the onset of diabetes mellitus after a pancreatectomy. The investigators will also monitor patients with pre-existing diabetes to see if their diabetes worsens or improves. Patients will be followed up to one year to track their diabetes status, postoperative outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pancreatectomy at our institution (e.g., pancreaticoduodenectomy, distal pancreatectomy, distal pancreatectomy and splenectomy, central pancreatectomy).

Exclusion Criteria:

* All patients who are on steroids or other medications whose potential side effects include development of diabetes mellitus or elevated blood glucose.
* Pregnant or nursing women.
* Patients with uncontrolled diabetes (HbA1c >8%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients scheduled to undergo a pancreatectomy for a pancreatic neoplasm
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Percent resected volume of pancreas and diabetes development | Postoperative up to one year

SECONDARY OUTCOMES:
QLQ-C30 Quality of Life Health Questionnaire | Postoperative up to one year
Blood glucose control | Postoperative up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rosemurgy, MD, Principal Investigator — Florida Hospital Tampa

IPD SHARING:
Plan to Share IPD: No